CLINICAL TRIAL: NCT02037412
Title: Impact of Ticagrelor on the Endothelial Healing Following Drug-eluting Stent Implantation in the Patients With Acute Coronary Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The patient registration was not successful.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0764
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2016-12

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction; Unstable Angina (Intermediate Coronary Syndrome)
Keywords: Ticagrelor; strut coverage; DES; ACS; OCT
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor Arm (Experimental): Ticagrelor Arm
  Interventions: Drug: Ticagrelor
- Clopidogrel Arm (Active Comparator): Clopidogrel Arm
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor - 180 mg loading and 90 mg bid maintenance for 3 months
  Arms: Ticagrelor Arm
Drug: Clopidogrel — Clopidogrel - 600 mg loading and 75 mg qd maintenance for 3 months
  Arms: Clopidogrel Arm

SUMMARY:
The investigators hypothesized that ticagrelor may enhance endothelial healing after DES implantation by increasing adenosine concentrations by the inhibition of adenosine uptake into erythrocytes, compared to clopidogrel. Thus, the investigators will evaluate the extent of endothelialization (stent strut coverage) and neointimal hyperplasia (neointimal thickness) 3 months after DES implantation by optical coherence tomography (OCT)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 20 years old
* Patients who are hospitalized and expected to undergo PCI for acute coronary syndrome, including acute myocardial infarction and unstable angina.

Exclusion Criteria:

* Age > 80 years
* Cardiogenic shock or unstable patients
* Increased risk of bleeding, anemia, thrombocytopenia
* A need for oral anticoagulation therapy
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Stent re-endothelialization | Three months after stent implantation
  Percentage of stent coverage measured by OCT
Neointimal hyperplasia | Three months after stent implantation
  Neointimal thickness measured by OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Patil SB, Jackman LE, Francis SE, Judge HM, Nylander S, Storey RF. Ticagrelor effectively and reversibly blocks murine platelet P2Y12-mediated thrombosis and demonstrates a requirement for sustained P2Y12 inhibition to prevent subsequent neointima. Arterioscler Thromb Vasc Biol. 2010 Dec;30(12):2385-91. doi: 10.1161/ATVBAHA.110.210732. Epub 2010 Nov 11. PMID 21071697
- [Background] Kim JS, Fan C, Choi D, Jang IK, Lee JM, Kim TH, Park SM, Paik SI, Ko YG, Hong MK, Jang Y, Chung N. Different patterns of neointimal coverage between acute coronary syndrome and stable angina after various types of drug-eluting stents implantation; 9-month follow-up optical coherence tomography study. Int J Cardiol. 2011 Feb 3;146(3):341-6. doi: 10.1016/j.ijcard.2009.07.012. Epub 2009 Aug 25. PMID 19709765